CLINICAL TRIAL: NCT07401953
Title: Long-term Fracture Risk in Living Kidney Donors
Brief Title: Fracture Risk in Living Kidney Donors
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021 0906 443 002
Record Dates: First submitted 2026-02-03; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Living Kidney Donor; Living Kidney Donation; Fractures; Nephrectomy,Kidney Donation; Fragility Fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Living kidney donor cohort: Living kidney donors who had a laparoscopic nephrectomy between July 1, 1992 and March 31, 2024, at transplant centres in the provinces of Ontario, Alberta, and British Columbia. Each nephrectomy date will serve as their cohort entry date.
  Interventions: Procedure: Nephrectomy
- Healthy non-donor cohort: A similarly healthy segment of the general provinical population selected using restriction and matching to emulate the health criteria required to be met for living kidney donation. We will randomly assign a cohort entry date (simulated nephrectomy date) to all residents in the province, according to the distribution of cohort-entry dates among donors (between July 1, 1992 and March 31, 2024).

INTERVENTIONS:
Procedure: Nephrectomy — Receipt of a nephrectomy for living kidney donation
  Groups: Living kidney donor cohort

SUMMARY:
We will conduct a population-based, matched retrospective cohort study using linked administrative healthcare databases from Ontario, Alberta, and British Columbia to evaluate the long-term risk of fractures among living kidney donors compared with a healthy cohort of nondonors. Living kidney donors who donated between 1992 and 2024 will be included and matched 1:10 to a carefully selected population of nondonors based on key demographic and clinical characteristics. The primary outcome is a composite of incident hip, femoral shaft, humeral, wrist/forearm, and pelvic fractures. Secondary outcomes will examine each fracture site separately. The results will provide evidence to inform clinical guidelines, support informed decision-making for potential donors and recipients, and guide counselling by transplant clinicians.

DETAILED DESCRIPTION:
* Summary *

Background: Individuals with chronic kidney disease have an increased risk of fracture, but the long-term fracture risk among living kidney donors remains unclear. Prior studies in donors have shown changes in bone biomarkers, including elevated levels of parathyroid hormone; however, follow-up has been limited (≤5 years), and these studies have not evaluated fracture outcomes. Only one prior study has assessed fracture risk in living kidney donors and found no increased risk, with up to 17 years of follow-up. Leveraging linked administrative healthcare data across three provinces, we can now evaluate fracture risk in living kidney donors with more than 25 years of follow-up and improve upon prior methodologies through rigorous matching strategies and control selection.

Methods: We will conduct a matched population-based retrospective cohort study of living kidney donors using provincial healthcare administrative databases from Ontario, Alberta, and British Columbia. Using linked databases from each province, we will identify individuals who have donated a kidney between 1992 and 2024 and compare them to matched nondonors (1:10) with similar baseline health status and demographic characteristics. Donors and nondonors will be matched at the time of donation for age, sex, year of nephrectomy (simulated nephrectomy in nondonors), residency (urban or rural), income quintile, and previous fracture. The primary outcome will be a composite measure of fragility fractures, including fractures of the hip, femur, humerus, wrist/forearm, and pelvis. Secondary outcomes will involve analyzing each of these fracture types separately. In a tertiary outcome analysis, we will examine vertebral fractures both as part of the composite fragility fracture outcome and independently, given the nature of how this fracture type is captured in health administrative data. Vertebral fractures are often underrecognized because they can be asymptomatic and may only be identified incidentally through imaging. We will use privacy-preserving methods to combine results and estimate risks across these three provinces, as individual-level data cannot be shared due to privacy constraints.

Study outcome: This study aims to determine whether living kidney donors have an increased risk of fragility fracture (defined as a composite of hip, femoral shaft, humeral, wrist/forearm, and pelvic fractures) compared with carefully selected nondonors of comparable baseline health. Secondary objectives include identifying risk factors for fracture in both donors and nondonors and evaluating fracture risk within prespecified subgroups.

* Literature Review *

Individuals with reduced kidney function, defined as an estimated glomerular filtration rate (eGFR) of 15-59 mL/min/1.73 m², have a 1.5- to 3-fold higher risk of fragility fractures compared with those with normal kidney function (eGFR ≥60 mL/min/1.73 m²) (Dooley et al., 2008; Dukas et al., 2005; Ensrud et al., 2007; Fried et al., 2007; Nickolas et al., 2006). Among living kidney donors, approximately 40% have an eGFR of 60-80 mL/min/1.73 m² and 10% have an eGFR of 30-59 mL/min/1.73 m² ten years post-donation (Garg et al., 2006; Ibrahim et al., 2006), raising concern about potential long-term skeletal consequences.

To date, only two studies have examined fracture risk in living kidney donors. A population-based matched retrospective cohort study by Garg and colleagues (2012), using ICES administrative data, found no significant difference in fracture risk between donors and nondonors after accounting for baseline health differences, with a maximum follow-up of 17 years. More recently, Kremers and colleagues (2024) used a survey-based approach and reported a lower overall fracture risk among donors but an increased risk of vertebral fractures compared with matched controls after a mean follow-up of 25 years. Together, these findings suggest that if an association between living kidney donation and fragility fractures exists, it may emerge over longer follow-up periods, particularly as donors age and kidney function declines below an eGFR of 60 mL/min/1.73 m². To ensure that living kidney donation remains safe across the donor lifespan, updated population-based analyses with extended follow-up and improved methodology are warranted.

* Research Setting *

The research will take place at ICES (ices.on.ca), a non-profit organization recognized under Ontario's health privacy legislation as a prescribed entity. This designation allows ICES to access and use health and demographic data without individual consent for the purpose of evaluating and improving the health system. The use of data in this project falls under Section 45 of Ontario's Personal Health Information Protection Act (PHIPA) and it does not require approval from a Research Ethics Board.

In Ontario, data will be obtained from several linked administrative databases, including the Trillium Gift of Life Network (TGLN), the Registered Persons Database (RPDB), the Ontario Health Insurance Plan (OHIP) database, and the Canadian Institute for Health Information (CIHI) Discharge Abstract Database (CIHI-DAD), National Ambulatory Care Reporting System (NACRS), and Same Day Surgery (SDS) databases. For most hospitalization and physician billing data, information is available from 1991 onward; therefore, July 1, 1992, will mark the start of the accrual period. We anticipate near-complete capture for all study variables. Living kidney donors will be identified primarily using TGLN, with CIHI-DAD used for donor identification in years where TGLN data are unavailable.

To ensure consistency across provinces, equivalent administrative databases will be used in Alberta and British Columbia. In Alberta, data will be accessed through the Alberta Kidney Disease Network (AKDN) and Alberta Health Services (AHS), subject to analyst assignment and data availability. Living kidney donors will be identified using CIHI-DAD. Demographic characteristics and vital statistics will be obtained from the Alberta Provincial Registry and Vital Statistics databases, while information on hospital admissions, diagnoses, and healthcare encounters will be drawn from CIHI-DAD, NACRS, and the Alberta Practitioner Claims database.

In British Columbia, data will be accessed through Population Data BC (PopDataBC) and the Healthcare Data Platform BC (HDPBC). Living kidney donors will be identified using the Patient Records and Outcome Management Information System (PROMIS) database, accessed through BC Renal. If data is unavailable, we will use CIHI-DAD to identify donors. Demographic and vital statistics data will be sourced from Population Data BC's Consolidation File/Central Demographics database. Hospital admissions, diagnoses, and health care visit data will be obtained from CIHI-DAD, CIHI-NACRS, and Population Data BC's Medical Services Plan database.

This retrospective cohort study will use existing administrative healthcare data. In accordance with best practices for observational research, the study description, design, and statistical analysis plan will be publicly registered on ClinicalTrials.gov prior to outcome analyses.

* Statistical Analysis *

Baseline characteristics: Continuous variables will be presented as mean (standard deviation) or median (interquartile range [IQR]), as appropriate, and categorical variables as frequency (percentage). Due to our large expected cohort size and the influence of sample size on statistical testing, the characteristics of donors and nondonors at the time of cohort entry will be compared prior to and after matching using standardized mean differences, where a value >0.10 is considered meaningfully different. Characteristics specific to the donors will also be reported depending on data availability (e.g., pre-nephrectomy kidney function and donor relationship to the recipient).

Period of observation: Participants will be accrued between July 1, 1992, and March 31, 2024, subject to data availability. Follow-up will begin at cohort entry and will be censored at the earliest occurrence of the relevant study outcome (time to first event), death, emigration from the province, or the end of the observation period (March 31, 2025).

Assessing risk of the primary, secondary, and tertiary outcomes: The primary analysis will evaluate the association between living kidney donation and the risk of hospitalization for a composite fragility fracture, defined as hip, femoral shaft, humeral, wrist/forearm, or pelvic fracture. Only the first fracture event will be considered. Hazard ratios (HRs) and 95% confidence intervals (CIs) will be estimated using Cox proportional hazards regression with robust variance estimation to account for correlation within matched sets. The proportional hazards assumption will be evaluated using a Kolmogorov-type supremum test based on 1,000 simulated patterns. If the proportional hazards assumption is violated, a stratified log-rank test will be used to assess statistical significance, and differences in restricted mean survival time at 20 years with corresponding 95% CIs will be reported. This analytical approach will be repeated for each fracture site examined separately (secondary outcomes: hip, femur, humerus, wrist/forearm, and pelvis) and for a composite outcome that additionally includes vertebral fractures and vertebral fractures separately (tertiary outcome).

Risk factor analysis: Risk factor analyses will be conducted to identify factors associated with fracture risk among living kidney donors and nondonors. Age, sex (male vs female), rurality of residence (urban vs rural), neighborhood income quintile (per quintile increase), year of donation (simulated donation in nondonors), and history of fracture within five years prior to cohort entry (yes vs no) will be examined as predictors of fracture risk. Associations will be estimated using Cox proportional hazards regression models, with results reported as hazard ratios and 95% confidence intervals.

Subgroup analysis: Prespecified subgroup analyses will be conducted to assess whether the association between living kidney donation and fracture risk varies across clinically relevant subgroups. Analyses will be stratified by age at cohort entry (<55 vs ≥55 years), sex (male vs female), and index period (1992-2001, 2002-2012, and 2013-2023). In addition, a combined age-sex subgroup will be examined using four categories (younger females, older females, younger males, and older males). For each subgroup, hazard ratios and 95% confidence intervals will be estimated using Cox proportional hazards regression with robust variance estimation, consistent with the primary analysis approach.

Combining outcome results from Ontario, Alberta and British Columbia: To improve statistical power and generalizability, results from Ontario, Alberta, and British Columbia will be combined for the outcomes. We will use a privacy-preserving Cox regression approach for multisite studies in which individual-level data cannot be shared (Shu et al., 2020). This method requires a single transfer of summary-level outputs from each province and yields results identical to those obtained from pooled individual-level data. The approach assumes province-specific baseline hazards and accommodates survival and binary outcomes, with confounding control (e.g., matching or weighting) conducted within each province. Summary-level risk-set tables generated by each province will be securely transferred to the coordinating site to estimate combined hazard or risk ratios with 95% confidence intervals. To comply with privacy regulations, all cell sizes of five or fewer will be suppressed (reported as ≤5) in publications, and all team members will adhere to required data confidentiality and data use agreements.

Additional prespecified analyses (Ontario only): We will conduct supplementary descriptive analyses in the Ontario cohort to characterize additional laboratory and medication variables related to bone health.

(i) We will report the number and proportion of individuals with multiple fractures during follow-up.

(ii) We will examine bone mineral density (BMD) testing, reporting the distribution of the number of tests during follow-up. These data reflect whether a test was performed, not the test results.

(iii) Among a sub-cohort aged ≥66 years at index, we will use the Ontario Drug Benefit (ODB) database to identify new osteoporosis-related prescriptions, excluding individuals with relevant prescriptions in the year prior to index to capture new users of these medications. Medications of interest include bisphosphonates, systemic estrogen/raloxifene, denosumab (after February 2012), prescription vitamin D/calcium, and teriparatide (after February 2006).

(iv) If an adequate amount of measurements is available in a sub-cohort, we will assess bone metabolism markers including parathyroid hormone, corrected calcium, alkaline phosphatase, 25-hydroxyvitamin D, and phosphate. Limitations related to laboratory data capture in our data sources may affect the completeness of follow-up test counts.

ELIGIBILITY:
*Donors* Inclusion Criteria: Living kidney donors who underwent donor nephrectomy in Ontario, Alberta, and British Columbia, Canada, between July 1, 1992, and March 31, 2024 are eligible to enter the study.

Exclusion criteria:

* We will exclude any person with data errors in their database records (such as missing or invalid age; we expect to exclude very few persons for these reasons). Data errors also include evidence of prior dialysis or a prior solid organ transplant, as such individuals are not eligible to become donors.
* We will exclude any person who was not a permanent resident of the province (i.e., they live outside of the province, and only came to the province to donate a kidney to their intended recipient). This will include anyone who is not eligible for the province's health insurance plan, anyone whose date of last contact in the databases is less than 1 year after the cohort entry date, and any person without a physician visit in the last 1-year.
* We will exclude any person who is <18 years of age on the date of nephrectomy (as only under exceptional circumstances should a person less than 18 be approved for living donation).

*Non-donors* Inclusion criteria: Before nephrectomy, living donors undergo rigorous health screening. We will select a similarly healthy segment of the general population using restriction and matching. We will randomly assign a cohort-entry date (simulated nephrectomy date) to all persons who were citizens in the province, according to the distribution of cohort-entry dates among donors (July 1, 1992, to March 31, 2024).

Exclusion Criteria:

* We will exclude any person with data errors in their database records (such as missing or invalid age).
* We will exclude any person who was not a permanent resident of the province. This will include anyone who is not eligible for the province's health insurance plan, anyone whose date of last contact in the databases is less than 1 year after the cohort entry date.
* We will exclude any person who is <18 years of age on the cohort entry date.
* We will exclude anyone who is pregnant at the time of index date.
* We will identify baseline illnesses and measures of healthcare access from historic records preceding the cohort entry date. We will then restrict the sample of eligible nondonors to persons without a recorded medical condition that could preclude donation. Such recorded medical conditions will include a hospitalization for mental illness in the prior year; an intensive care unit admission in the prior year; a hospitalization for palliative care services in the prior year; multiple hospital admissions in the prior year; high comorbidity (as assessed by the Charlson comorbidity index and adjusted clinical group scores); receipt of home oxygen therapy; residence at a long-term care facility; dementia; any record of prior nephrology consultation or kidney disease (including receipt of dialysis, a kidney biopsy, or a kidney procedure such as a partial or complete nephrectomy); previous solid organ transplant; disorders of the kidneys, ureters, or bladder; any record of cardiovascular disease (congestive heart failure, cardiovascular procedures, myocardial infarction, peripheral vascular disease, abdominal aortic aneurysm repair, ischemic stroke); hypertension in individuals <50 years of age (persons with this condition are not accepted as donors in Ontario); any record of obstructive sleep apnea; any cancer diagnosis; any liver disease or cirrhosis; diabetes; any serious infection (hepatitis, HIV, infective endocarditis); any record of autoimmune rheumatic conditions (such as rheumatoid arthritis or systemic lupus erythematosus); and any record of alcoholism.
* To ensure the nondonors have the same opportunity as donors to obtain health care services from physicians, we will exclude nondonors who had no evidence of a family physician visit in the 2 years prior to index. We will also exclude nondonors with more than 5 family physician visits in the 2 years prior to index, as this could suggest they have an active health issue that needs attention before they would proceed to donate.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Living kidney donors matched to nondonors from the general population with similar indicators of baseline health.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Actual)
Dates: Start 1992-07-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Fragility fracture | Donors and their matched non-donors will enter the cohort between July 1, 1992 and March 31, 2023, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2024).
  Hospital admission, emergency department visit, and/or billing receipt for a fragility fractures, defined as a composite of hip, femur, humerus, wrist/forearm, and pelvis.

SECONDARY OUTCOMES:
Each fragility fracture type/location | Donors and their matched non-donors will enter the cohort between July 1, 1992 and March 31, 2023, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2024).
  Hospital admission, emergency department visit, and/or billing receipt for first event of each type of fragility fracture, hip, femur, humerus, wrist/forearm, or pelvis.

OTHER OUTCOMES:
Spinal/vertebral fragility fractures | Donors and their matched non-donors will enter the cohort between July 1, 1992 and March 31, 2023, and will be followed until study outcome (first event), death, emigration from the province, or the end of the observation period (March 31, 2024).
  Hospital admission, emergency department visit, and/or billing receipt for a fragility fracture, defined as a composite of hip, femur, humerus, wrist/forearm, pelvis, and clinical spinal/vertebral. And hospital admission, emergency department visit, and/or billing receipt for first event of clinical spinal/vertebral fracture.

IPD SHARING:
Plan to Share IPD: No
The dataset from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). Similarly, the Alberta and British Columbia datasets are held securely by their respective data stewards, and access is governed by provincial privacy legislation and data sharing agreements. The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Garg AX, Pouget J, Young A, Huang A, Boudville N, Hodsman A, Adachi JD, Leslie WD, Cadarette SM, Lok CE, Monroy-Cuadros M, Prasad GV, Thomas SM, Naylor K, Treleavan D; Donor Nephrectomy Outcomes Research (DONOR) Network. Fracture risk in living kidney donors: a matched cohort study. Am J Kidney Dis. 2012 Jun;59(6):770-6. doi: 10.1053/j.ajkd.2012.01.013. Epub 2012 Apr 1. PMID 22472209
- [Background] Nickolas TL, McMahon DJ, Shane E. Relationship between moderate to severe kidney disease and hip fracture in the United States. J Am Soc Nephrol. 2006 Nov;17(11):3223-32. doi: 10.1681/ASN.2005111194. Epub 2006 Sep 27. PMID 17005938
- [Background] Ibrahim HN, Rogers T, Tello A, Matas A. The performance of three serum creatinine-based formulas in estimating GFR in former kidney donors. Am J Transplant. 2006 Jun;6(6):1479-85. doi: 10.1111/j.1600-6143.2006.01335.x. PMID 16686774
- [Background] Garg AX, Muirhead N, Knoll G, Yang RC, Prasad GV, Thiessen-Philbrook H, Rosas-Arellano MP, Housawi A, Boudville N; Donor Nephrectomy Outcomes Research (DONOR) Network. Proteinuria and reduced kidney function in living kidney donors: A systematic review, meta-analysis, and meta-regression. Kidney Int. 2006 Nov;70(10):1801-10. doi: 10.1038/sj.ki.5001819. Epub 2006 Sep 27. PMID 17003822
- [Background] Fried LF, Biggs ML, Shlipak MG, Seliger S, Kestenbaum B, Stehman-Breen C, Sarnak M, Siscovick D, Harris T, Cauley J, Newman AB, Robbins J. Association of kidney function with incident hip fracture in older adults. J Am Soc Nephrol. 2007 Jan;18(1):282-6. doi: 10.1681/ASN.2006050546. Epub 2006 Dec 13. PMID 17167115
- [Background] Ensrud KE, Lui LY, Taylor BC, Ishani A, Shlipak MG, Stone KL, Cauley JA, Jamal SA, Antoniucci DM, Cummings SR; Osteoporotic Fractures Research Group. Renal function and risk of hip and vertebral fractures in older women. Arch Intern Med. 2007 Jan 22;167(2):133-9. doi: 10.1001/archinte.167.2.133. PMID 17242313
- [Background] Dukas L, Schacht E, Stahelin HB. In elderly men and women treated for osteoporosis a low creatinine clearance of <65 ml/min is a risk factor for falls and fractures. Osteoporos Int. 2005 Dec;16(12):1683-90. doi: 10.1007/s00198-005-1903-7. Epub 2005 Jun 3. PMID 15933802
- [Background] Dooley AC, Weiss NS, Kestenbaum B. Increased risk of hip fracture among men with CKD. Am J Kidney Dis. 2008 Jan;51(1):38-44. doi: 10.1053/j.ajkd.2007.08.019. PMID 18155531